# Examining Peer Influences in Alcohol and Sexual Violence among Marines Using a Dyadic Multimethod Approach

**NCT Number TBD** 

November 20, 2025

# Georgia State University Informed Consent

Title: Military Dyadic Study

Principal Investigator: Amanda K. Gilmore, PhD

**Sponsor:** National Institute on Alcohol Abuse and Alcoholism

#### **Introduction and Key Information**

• You are invited to take part in a research study. It is up to you to decide to participate.

- The purpose of this study is to understand alcohol use, entertainment habits and preferences, and social behavior of men currently serving in the United States Marine Corps (USMC).
- Your role in the study will last about 4 hours over two weeks. You will be asked to complete a:
  - o 20-minute online orientation with a member of the research team
  - 30-minute online survey about alcohol, entertainment habits and preferences, and social behavior
  - two brief online surveys a day for 14 days that take 5 minutes each. You will respond once in the morning and once in the evening at a time you choose. You will also be asked to respond when you are drinking. You will be asked about your current and recent thoughts and behaviors.
  - 30-minute online session with your friend, another pair of Marines, and up to two
    members of the research team. The session will take place on video (e.g., Zoom) and
    you will be asked to do an entertainment task.
- Risks include possible discomfort when asked to answer sensitive questions, including questions about your sexual experiences and potentially traumatic experiences during deployment. You could also be uncomfortable when reading about a film clip with sexual content, or from having to choose which film clip to show the other person.
- This study is not designed to benefit you. Overall, we hope to better understand alcohol, entertainment habits and preferences, and social behavior of men in the USMC.

### Purpose

The goal of this study is to learn about the drinking habits, entertainment choices, and social behavior of men who are in the USMC. You are invited to participate because you are a man aged 21 or older who drinks alcohol and you are currently serving in the U.S. Marine Corps. You must be able and willing to recruit a fellow man in the USMC. This man should be someone who you have consumed alcohol with at least twice in the past month. A total of 326 people will be invited to take part in this study.

#### **Procedures**

This study will last 2 weeks. You will be asked to complete the following:

A 20-minute one-on-one orientation via Zoom with a member of the research team

Version Date: 11-20-2025

- A 30-minute online survey about alcohol, your entertainment habits and preferences, and social behavior. Your partner in the research will also provide information about their perceptions of your drinking and behavior in the questionnaire.
- Two brief online surveys a day for 14 days. You will respond once in the morning and once in the evening at a time you choose. You will also be asked to respond when you are drinking. You will be asked about your current and recent thoughts and behaviors. These are called EMA reports.
- A 30-minute online session on Zoom. The session will include your research partner, another
  pair of Marines, and up to two members of the research team. An additional member of the
  research team may observe for training purposes. Four minutes of the Zoom session will be
  recorded for quality control.

#### **Future Research**

Researchers will remove identifying information and may use your data for future research. If we do this, we will not ask for any additional consent from you.

### Risks

You may feel some discomfort when asked to answer questions about sensitive information, including questions about your sexual experiences and potentially traumatic experiences during deployment. You may also be uncomfortable when reading about a film clip with sexual content or from having to choose which film clip to show the other person.

No injury is expected from this study. If you believe you have been harmed, contact the research team as soon as possible. Georgia State University and the research team have not set aside funds to compensate for any injury.

### **Benefits**

This study is not designed to benefit you. Overall, we hope to better understand alcohol, entertainment habits and preferences, and social behavior of men currently serving in the USMC.

### **Alternatives**

The alternative to taking part in this study is to not take part in the study.

#### Compensation

You will be paid \$40 for the baseline survey and \$40 for the Orientation Session. You will also be paid \$10 per completed scheduled EMA report ( $$10 \times 2$ times per day x 14 days = $280$ ), and a \$5 bonus for each week in which 80% or more of scheduled EMA reports are completed ( $$5 \times 2$ weeks = $10$ ). You will be paid \$80 for the online experiment session. You may receive up to \$450 total. If you withdraw from the study, you will be paid for the time you were in the study. Payments will be in the form of an Amazon gift card.

### **Voluntary Participation and Withdrawal**

Version Date: 11-20-2025

You do not have to be in this study. If you decide to participate and change your mind, you have the right to drop out at any time. You may skip questions or stop participating at any time.

# Confidentiality

We will keep your records private to the extent allowed by law. The following people and entities will have access to the data:

- Amanda K. Gilmore and approved research staff
- GSU Institutional Review Board
- Office for Human Research Protection (OHRP)
- National Institute on Alcohol Abuse and Alcoholism

Deidentified data from this study will also be submitted to the National Institute on Alcohol Abuse and Alcoholism Database (NIAAADA) at the National Institutes of Health (NIH). Deidentified data means that all personal information about you (such as name, address, birth date and phone number) is removed and replaced with a number. Other researchers will be able to request access to the data; however, your identifying information will not be connected to the data, and anyone with access to the data must promise to keep your data safe, and they must not to try to learn your identity. Although researchers and NIH will make every attempt to protect your identity, your data could be accidentally shared with someone without approval who may attempt to learn your identity.

You may decide now or later that you do not want your deidentified data to be added to the NIAAADA. You can still take part in this research study even if you decide that you do not want your data to be added to the NIAAADA. If you know now that you do not want your data in the NIAAADA, you may opt out on the next page. If you decide any time after today that you do not want your data to be added to the NIAAADA, please call or email the study staff. They will tell NIAAADA to stop sharing your data. Once your data is part of the NIAAADA, the study researchers cannot take back the data that was shared before they were notified that you changed your mind. For more information about NIAAADA, visit <a href="https://nda.nih.gov/niaaa">https://nda.nih.gov/niaaa</a>.

We will use a study number rather than your name on study records. All information will be stored on secure online website. The code sheet linking your information to the study number will be stored in a password protected file on a secure online website while you are in the study. We will destroy the code sheet after you have finished the study. The audio recordings will be transcribed. We will remove any identifying information from the transcripts. After the study, the recordings will be destroyed. When we present or publish the results of this study, we will not use your name or other information that may identify you.

To help us protect your privacy, we have a Certificate of Confidentiality from the National Institutes of Health (NIH). With this Certificate, we can't be forced by a court order or subpoena to disclose information that could identify you in any civil, criminal, administrative, legislative or other proceeding.

There are circumstances where the Certificate doesn't protect against disclosure of your personally identifiable information:

When the US government is inspecting or evaluating federally-funded studies

- When information must be disclosed to meet FDA requirements
- If you give someone written permission to receive research information or you voluntarily disclose your study information
- If the researcher reports that you threatened to harm yourself or others
- In cases of child abuse reported by the researcher
- If the investigator reports cases of contagious disease (such as HIV) to the state

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## **Contact Information**

Contact Amanda K. Gilmore, PhD at militaryresearch@gsu.edu:

- If you have questions about the study or your part in it
- If you have questions, concerns, or complaints about the study

The IRB at Georgia State University reviews all research that involves human participants. You can contact the IRB if you would like to speak to someone who is not involved directly with the study. You can contact the IRB with concerns, problems, information, input, or questions about your rights as a research participant. Contact the IRB at 404-413-3500 or <a href="mailto:irb@gsu.edu">irb@gsu.edu</a>.

# **Consent**

You can print or save a copy of the form for your records.

If you are willing to volunteer for this research, please click "agree" below to continue.

- I agree to participate, continue to the study
- I do not agree to participate, do not continue to the study

Version Date: 11-20-2025